CLINICAL TRIAL: NCT03992872
Title: A Phase 2 Open-label Study to Assess the Safety and Immunogenicity of an Alum-adjuvanted Chikungunya Virus-like Particle Vaccine (PXVX0317) in Prior Recipients of Other Alphavirus Vaccines Versus Alphavirus Naïve Controls.
Brief Title: Phase 2 Open-label Study of Alum-adjuvanted Chikungunya Virus-like Particle Vaccine (PXVX0317)
Acronym: WRAIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EBSI-CV-317-002
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Chikungunya
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Intervention Model Description: Open Label Safety and Immunogenicity
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prior Alpha (Experimental): All study participants received the same Investigational Product according to the same schedule. Participants were prior recipients of experimental alphavirus vaccines.
  Interventions: Biological: Chikungunya
- Control: Naïve Alpha (Active Comparator): All study participants received the same Investigational Product according to the same schedule. The alphavirus vaccine naïve participants will serve as controls for determining the effect of pre-existing alphavirus immunity on vaccine safety and immunogenicity.
  Interventions: Biological: Chikungunya

INTERVENTIONS:
Biological: Chikungunya — Virus Like Particle

SUMMARY:
This was a phase 2 parallel-group age- and gender-matched open label study in healthy adults 18-65 years of age to assess the safety and immunogenicity of an alum-adjuvanted chikungunya virus-like particle vaccine (PXVX0317; CHIKV VLP vaccine) in prior recipients of other alphavirus vaccines versus alphavirus naïve controls.

DETAILED DESCRIPTION:
It is currently unknown whether prior exposure to heterologous alphaviruses will enhance or interfere with immune responses to chikungunya virus (CHIKV) exposure or vaccination. The objective of this study was to evaluate the safety and immunogenicity of the chikungunya vaccine candidate PXVX0317 when administered to prior recipients of experimental alphavirus vaccines versus alphavirus naïve gender- and age-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old (inclusive)
* For women of childbearing potential, a negative pregnancy test at screening and on vaccination day, practicing highly effective contraception for at least 30 days prior to vaccination, and willing to use a highly effective method of contraception through study completion.
* Able and willing to provide informed consent for study participation prior to screening procedures.
* Free of obvious health problems as established by medical history and clinical examination at screening and enrollment.
* Available to participate for the duration of the study (approximately 8 months).
* For the cohort of prior alphavirus vaccine recipients, a documented history of prior alphavirus vaccination.

Exclusion Criteria:

* Acute disease or febrile illness at the time of screening or enrollment.
* Clinically significant cardiac, respiratory, rheumatologic or other medical or psychiatric condition that, in the opinion of the Investigator, places the subject at increased risk or affects their ability to understand and comply with study procedures.
* Abnormal screening lab test result that, in the opinion of the investigator, obscures interpretation of the safety data or suggests a clinically significant cardiac, respiratory, rheumatologic or other medical condition that places the subject at increased risk.
* Pregnant, lactating or planning to become pregnant during the study period.
* Laboratory evidence of infection with Hepatitis B, C or HIV.
* History of naturally (non-laboratory) acquired chikungunya or other alphavirus infection or travel to a WHO-designated chikungunya-endemic region within 30 days prior to Day 1.
* History of acute allergic reaction to any component of CHIKV VLP vaccine or Alhydrogel®.
* Current (30 days prior to Day 1) or anticipated use of systemic immunomodulatory or immunosuppressive medications.
* History of splenectomy, immunosuppressive condition, autoimmune disease, or immunodeficient condition.
* Family history of congenital or hereditary immunodeficiency.
* Suspected or known current alcohol abuse that, in the opinion of the Investigator, would interfere with the subject's ability to understand and comply with study procedures.
* Current intravenous drug use.
* Prior receipt of an investigational chikungunya vaccine.
* Receipt or planned receipt of any licensed vaccine from 30 days prior to Day 1 through Day 29 study visit.
* Participation in another clinical trial during the study period in which an investigational product is administered.
* For the alphavirus naïve group, history of prior alphavirus vaccination is exclusionary.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McCarty, MD, Study Director — Emergent BioSolutions
Locations (2):
- United States (2):
  - United States Army Medical Research Institute of Infectious Diseases, Fort Deterick, Maryland
  - Walter Reed Army Institute of Research, Silver Spring, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamer MJ, McCarty JM, Pierson BC, Regules JA, Mendy J, Sanborn AD, Gardner CL, Haller JM, Gregory MK, Liggett DL, Glass PJ, Ghosh N, Royalty Tredo S, Warfield KL, Burke CW, Lee C, Saunders D, Bedell L, Richardson JS. Safety and immunogenicity of an adjuvanted chikungunya virus virus-like particle (CHIKV VLP) vaccine in previous recipients of other alphavirus vaccines versus alphavirus vaccine-naive controls: an open-label, parallel-group, age-matched, sex-matched, phase 2 randomised controlled study. Lancet Microbe. 2025 Apr;6(4):101000. doi: 10.1016/j.lanmic.2024.101000. Epub 2025 Feb 12. PMID 39954701

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two US sites, Walter Reed Army Institute of Research (WRAIR) Clinical Trials Center (CTC) and US Army Medical Research Institute for Infectious Disease (USAMRIID) immunization clinic.
Groups:
- Experimental : Prior Alpha: All study participants received the same Investigational Product according to the same schedule. Subjects were prior recipients of experimental alphavirus vaccines.
- Control: Naive Alpha: All study participants received the same Investigational Product according to the same schedule. The alphavirus vaccine naïve subjects served as controls.
Period: Overall Study
Arm/Group | Experimental : Prior Alpha | Control: Naive Alpha
Started | 30 | 30
Exposed (Screened subjects who received study vaccination.) | 30 | 30
Safety (Subjects who received study vaccination and provided safety assessment data.) | 30 | 30
mITT (Exposed subjects who had evaluable results from both Day 1 and at least one later on-study sample.) | 30 | 30
Immunogenicity Evaluable (Exposed subjects who met the IEP criteria as detailed in the SAP.) | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Naive Alpha: All study participants received the same Investigational Product according to the same schedule. The alphavirus vaccine naïve subjects serves as controls.
- Total: Total of all reporting groups
Arm/Group | Experimental : Prior Alpha | Control: Naive Alpha | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 20 | 20 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 28 | 29 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 12 | 14
  White | 26 | 14 | 40
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 171.12 (11.37) | 175.10 (11.16) | 173.11 (11.35)
Weight [Mean (Standard Deviation); unit: Kg] | 90.99 (19.19) | 94.64 (18.14) | 92.82 (18.60)
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 31.04 (6.11) | 30.78 (4.72) | 30.91 (5.42)
Time Since Prior Alphavirus Vaccine [Mean (Standard Deviation); unit: years] | 16.2 (8.3) | NA (NA) — Applies only to subjects in the Prior Alpha arm. | 16.2 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 4-fold Rise in Anti-CHIKV Neutralizing Antibody Response
Description: Seroconversion, defined as a 4-fold or greater rise in neutralizing antibody against chikungunya virus, as determined by luciferase-based assay (NT80), induced by PXVX0317.
  PXVX0317 was administered to prior alphavirus vaccine recipients versus gender- and age-matched controls.
Time Frame: Day 22 (21 days after vaccination)
Population: Immunogenicity evaluable population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Experimental: Prior Alpha: All study participants received the same Investigational Product according to the same schedule. Participants were prior recipients of experimental alphavirus vaccines.
- Control: Naive Alpha: All study participants received the same Investigational Product according to the same schedule. The alphavirus vaccine naïve participants serve as controls.
Arm/Group | Experimental: Prior Alpha | Control: Naive Alpha
Number analyzed (Participants) | 30 | 30
percentage of participants | 100 [88.6 to 100] | 100 [88.6 to 100]
Statistical Analysis 1: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Test type: Superiority — The significance of the difference between groups in seroconversion rates was assessed using a Fisher's exact test. The percentage who seroconverted in each group was presented along with its 95% CI calculated using the Wilson method. The Newcombe method was use to estimate the 95% confidence interval for the difference between groups in the percentage of subjects who seroconverted; p = 1, Fisher Exact; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-11.4 to 11.4]

2. Secondary Outcome: Geometric Mean Titer of Anti-CHIKV Neutralizing Antibody Response
Description: Evaluation of Geometric Mean Titer of Anti-CHIKV neutralizing antibodies, determined by luciferase-based assay (NT80), in prior alphavirus vaccine recipients versus alphavirus-naïve controls.
Time Frame: Day 1, 8, 22, 29, 57, 182
Population: Immunogenicity evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Experimental: Prior Alpha | Control: Naive Alpha
Number analyzed (Participants) | 30 | 30
titers
  Day 1 | 9.21 [7.80 to 10.87] | 7.69 [NA to NA] — Not estimable due to lack of response; all baseline values in this group were < the limit of detection (LOD) (15) and imputed as LOD/2.
  Day 8 | 271.88 [163.72 to 451.49] | 87.48 [52.66 to 145.30]
  Day 22 | 2032.45 [1412.95 to 2923.56] | 2299.18 [1598.09 to 3307.84]
  Day 29 | 1555.60 [1081.46 to 2237.61] | 1772.54 [1118.75 to 2808.39]
  Day 57 | 727.91 [540.94 to 979.52] | 814.64 [567.46 to 1169.49]
  Day 182 | 294.35 [207.45 to 417.66] | 328.89 [231.75 to 466.74]
Statistical Analysis 1: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 1: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; P- value = NE (Not estimable due to lack of response; all baseline values in this group were <LOD and imputed as LOD/2, or 7.5); P-values were based on an ANOVA model with log10-transformed titer as the dependent variable and study arm, age, and gender as predictors; GMR (Prior Alpha / Naïve Alpha) = 1.20 — Differences in least squares means from the ANOVA model were back-transformed and reported as geometric mean ratios with 95% confidence intervals. 95% CI [NE,NE] NE = Not estimable due to lack of response
Statistical Analysis 2: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 8: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; p = 0.0019, ANOVA; [statistical method as in outcome 2, analysis 1]; GMR (Prior Alpha / Naïve Alpha) = 3.11, 95% CI 2-sided [1.55 to 6.23] — Differences in least squares means from the ANOVA model were back-transformed and reported as geometric mean ratios with 95% confidence intervals
Statistical Analysis 3: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 22: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; p = 0.6223, ANOVA; [statistical method as in outcome 2, analysis 1]; GMR (Prior Alpha / Naïve Alpha) = 0.88, 95% CI 2-sided [0.54 to 1.46] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 4: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 29: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; p = 0.6444, ANOVA — P-values were based on an ANOVA model with log10-transformed titer as the dependent variable and study arm, age, and gender as predictors; GMR (Prior Alpha / Naïve Alpha) = 0.88, 95% CI 2-sided [0.50 to 1.55] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 5: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 57: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; p = 0.6198, ANOVA — [p-value comment as in outcome 2, analysis 4]; GMR (Prior Alpha / Naïve Alpha) = 0.89, 95% CI 2-sided [0.57 to 1.41] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 6: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 182: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; p = 0.6451, ANOVA — [p-value comment as in outcome 2, analysis 4]; GMR (Prior Alpha / Naïve Alpha) = 0.89, 95% CI 2-sided [0.55 to 1.45] — [estimate comment as in outcome 2, analysis 2]

3. Secondary Outcome: Percentage of Participants With 4-fold Rise in Anti-CHIKV Neutralizing Antibody Response
Description: Evaluation of seroconversion rate of Anti-CHIKV neutralizing antibodies, determined by luciferase-based assay (NT80), in prior alphavirus vaccine recipients versus alphavirus-naïve controls.
Time Frame: Day 8, 29, 57, 182
Population: Immunogenicity evaluable population.
  11 alphavirus naïve subjects were unable to attend their scheduled visit at Day 29; 10 of those subjects also missed their Day 57 visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Prior Alpha | Control: Naive Alpha
Number analyzed (Participants) | 30 | 30
percentage of participants
  Day 8 | 93.3 [78.7 to 98.2] | 66.7 [48.8 to 80.8]
  Day 29: number analyzed (Participants) | 30 | 19
  Day 29 | 100 [88.6 to 100] | 100 [83.2 to 100]
  Day 57: number analyzed (Participants) | 30 | 20
  Day 57 | 100 [88.6 to 100] | 100 [83.9 to 100]
  Day 182 | 86.7 [70.3 to 94.7] | 100 [88.6 to 100]
Statistical Analysis 1: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Test type: Superiority; p = 0.0211, Fisher Exact; Day 8 Note: A subject has a 4-fold rise at a visit if they achieve a titer at that visit that is at least 4-fold higher than their Day 1 titer
Statistical Analysis 2: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Test type: Superiority; p = 1.0000, Fisher Exact; Day 29. Note: A subject has a 4-fold rise at a visit if they achieve a titer at that visit that is at least 4-fold higher than their Day 1 titer
Statistical Analysis 3: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Test type: Superiority; p = 1.0000, Fisher Exact; Day 57. Note: A subject has a 4-fold rise at a visit if they achieve a titer at that visit that is at least 4-fold higher than their Day 1 titer
Statistical Analysis 4: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Test type: Superiority; p = 0.1124, Fisher Exact; Day 182. Note: A subject has a 4-fold rise at a visit if they achieve a titer at that visit that is at least 4-fold higher than their Day 1 titer

4. Secondary Outcome: Percentage of Participants With Anti-CHIKV Neutralizing Antibody at or Above Selected Thresholds
Description: Evaluation of Anti-CHIKV neutralizing antibody response, as determined by luciferase-based assay (NT80), via proportion of participants with titers of at least 40, 160 or 640 on Days 1, 8, 22, 29, 57 and 182.
Time Frame: Day 1, 8, 22, 29, 57, 182
Population: Immunogenicity evaluable population. 11 alphavirus naïve participants were unable to attend their scheduled visit at Day 29; 10 of those participants also missed their Day 57 visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Prior Alpha | Control: Naive Alpha
Number analyzed (Participants) | 30 | 30
percentage of participants
  Day 1 (Titer >=40) | 3.3 [0.6 to 16.7] | 0 [0.0 to 11.4]
  Day 1 (Titer >=160) | 3.3 [0.6 to 16.7] | 0 [0.0 to 11.4]
  Day 1 (Titer >=640) | 0 [0.0 to 11.4] | 0 [0.0 to 11.4]
  Day 8 (Titer >=40) | 96.7 [83.3 to 99.4] | 73.3 [55.6 to 85.8]
  Day 8 (Titer >=160) | 70.0 [52.1 to 83.3] | 40 [24.6 to 57.7]
  Day 8 (Titer >=640) | 26.7 [14.2 to 44.4] | 10.0 [3.5 to 25.6]
  Day 22 (Titer >=40) | 100 [88.6 to 100] | 100 [88.6 to 100]
  Day 22 (Titer >=160) | 100 [88.6 to 100] | 100 [88.6 to 100]
  Day 22 (Titer >=640) | 73.3 [55.6 to 85.8] | 93.3 [78.7 to 98.2]
  Day 29 (Titer >=40): number analyzed (Participants) | 30 | 19
  Day 29 (Titer >=40) | 100 [88.6 to 100] | 100 [83.2 to 100]
  Day 29 (Titer >=160): number analyzed (Participants) | 30 | 19
  Day 29 (Titer >=160) | 100 [88.6 to 100] | 100 [83.2 to 100]
  Day 29 (Titer >=640): number analyzed (Participants) | 30 | 19
  Day 29 (Titer >=640) | 76.7 [59.1 to 88.2] | 94.7 [75.4 to 99.1]
  Day 57 (Titer >=40): number analyzed (Participants) | 30 | 20
  Day 57 (Titer >=40) | 100 [88.6 to 100] | 100 [83.9 to 100]
  Day 57 (Titer >=160): number analyzed (Participants) | 30 | 20
  Day 57 (Titer >=160) | 90.0 [74.4 to 96.5] | 95 [76.4 to 99.1]
  Day 57 (Titer >=640): number analyzed (Participants) | 30 | 20
  Day 57 (Titer >=640) | 63.3 [45.5 to 78.1] | 75 [53.1 to 88.8]
  Day 182 (Titer >=40) | 93.3 [78.7 to 98.2] | 100 [88.6 to 100]
  Day 182 (Titer >=160) | 76.7 [59.1 to 88.2] | 76.7 [59.1 to 88.2]
  Day 182 (Titer >=640) | 20.0 [9.5 to 37.3] | 30.0 [16.7 to 47.9]
Statistical Analysis 1: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 1 : Subjects with Titer >=40; Test type: Superiority; p > 0.9999, Fisher Exact
Statistical Analysis 2: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point Day 1: Subjects with Titer >=160; Test type: Superiority; p > 0.9999, Fisher Exact
Statistical Analysis 3: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 1: Subjects with Titer >=640; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 4: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 8 : Subjects with Titer >=40; Test type: Superiority; p = 0.0257, Fisher Exact
Statistical Analysis 5: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point Day 8: Subjects with Titer >=160; Test type: Superiority; p = 0.0370, Fisher Exact
Statistical Analysis 6: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 8: Subjects with Titer >=640; Test type: Superiority; p = 0.1806, Fisher Exact
Statistical Analysis 7: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 22: Subjects with Titer >=40; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 8: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point Day 22: Subjects with Titer >=160; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 9: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point Day 22: Subjects with Titer >=640; Test type: Superiority; p = 0.0797, Fisher Exact
Statistical Analysis 10: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 29: Subject with Titer >=40; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 11: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 29: Subject with Titer >=160; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 12: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 29: Subject with Titer >= 640; Test type: Superiority; p = 0.1284, Fisher Exact
Statistical Analysis 13: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 57: Subject with Titer >= 40; Test type: Superiority; p = 1.0000, Fisher Exact
Statistical Analysis 14: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 57: Subject with Titer>=160; Test type: Superiority; p = 0.6411, Fisher Exact
Statistical Analysis 15: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 57: Subject with Titer>=640; Test type: Superiority; p = 0.5382, Fisher Exact
Statistical Analysis 16: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 182: Subject with Titer >= 40; Test type: Superiority; p = 0.4915, Fisher Exact
Statistical Analysis 17: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 182: Subject with Titer >= 160; Test type: Superiority; p > 0.9999, Fisher Exact
Statistical Analysis 18: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-Chikungunya neutralizing activity at or above selected thresholds by time point. Day 182: Subject with Titer >= 640; Test type: Superiority; p = 0.5520, Fisher Exact

5. Secondary Outcome: Geometric Mean Titer of Anti-CHIKV Total Antibody Response
Description: Evaluation of Geometric Mean Titer of Anti-CHIKV total antibodies, determined by immunoassay (ELISA), in prior alphavirus vaccine recipients versus alphavirus-naïve controls.
Time Frame: Day 1, 22, 29
Population: Immunogenicity evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Experimental: Prior Alpha | Control: Naive Alpha
Number analyzed (Participants) | 30 | 30
titers
  Day 1 | 39.03 [29.85 to 51.03] | 25.77 [19.71 to 33.70]
  Day 22 | 2451.60 [1770.49 to 3394.72] | 1338.90 [966.77 to 1854.27]
  Day 29: number analyzed (Participants) | 30 | 19
  Day 29 | 2010.72 [1444.72 to 2798.46] | 1194.75 [786.21 to 1815.57]
Statistical Analysis 1: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 1: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; p = 0.0277, ANOVA — [p-value comment as in outcome 2, analysis 4]; GMR (Prior Alpha / Naïve Alpha) = 1.51, 95% CI 2-sided [1.05 to 2.19] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 22: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; p = 0.0088, ANOVA — [p-value comment as in outcome 2, analysis 4]; GMR (Prior Alpha / Naïve Alpha) = 1.83, 95% CI 2-sided [1.17 to 2.86] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 29: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; p = 0.0475, ANOVA — [p-value comment as in outcome 2, analysis 4]; GMR (Prior Alpha / Naïve Alpha) = 1.68, 95% CI 2-sided [1.01 to 2.82] — [estimate comment as in outcome 2, analysis 2]

6. Secondary Outcome: Percentage of Participants With 4-fold Rise in Anti-CHIKV Total Antibody Response
Description: Evaluation of seroconversion rate of Anti-CHIKV total antibodies, determined by immunoassay, on Days 22 and 29, where seroconversion was a 4-fold rise in titer over baseline.
Time Frame: Day 22, 29
Population: Immunogenicity evaluable population. 11 alphavirus naïve participants were unable to attend their scheduled visit at Day 29.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Prior Alpha | Control: Naive Alpha
Number analyzed (Participants) | 30 | 30
percentage of participants
  Day 22 | 100 [88.6 to 100] | 100 [86.6 to 100]
  Day 29: number analyzed (Participants) | 30 | 19
  Day 29 | 100 [88.6 to 100] | 100 [83.2 to 100]
Statistical Analysis 1: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Test type: Superiority; p = 1.00, Fisher Exact; Day 22. Note: A subject has a 4-fold rise at a visit if they achieve a titer at that visit that is at least 4-fold higher than their Day 1 titer
Statistical Analysis 2: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Test type: Superiority; p = 1.00, Fisher Exact; [statistical method as in outcome 3, analysis 2]

7. Secondary Outcome: Geometric Mean Titer of Anti-VEEV Neutralizing Antibody Response
Description: Evaluation of Geometric Mean Titer of Anti-VEEV neutralizing antibodies, determined by Plaque-Reduction Neutralization Test (PRNT80), in prior alphavirus vaccine recipients versus alphavirus-naïve controls
Time Frame: Day 1, 22, 29
Population: Immunogenicity evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Experimental: Prior Alpha | Control: Naive Alpha
Number analyzed (Participants) | 30 | 30
titers
  Day 1 | 449.82 [262.84 to 769.80] | 9.96 [NA to NA] — Not estimable due to lack of response
  Day 22 | 467.95 [278.47 to 786.34] | 9.89 [NA to NA] — Not estimable due to lack of response
  Day 29: number analyzed (Participants) | 30 | 19
  Day 29 | 538.63 [291.97 to 993.67] | 9.66 [NA to NA] — Not estimable due to lack of response
Statistical Analysis 1: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 1: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; P-values were based on an ANOVA model with log10-transformed titer as the dependent variable and study arm, age, and gender as predictors. P-value = NE NE = Not estimable due to lack of response; GMR (Prior Alpha / Naïve Alpha) = 45.17 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 22: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; [p-value comment as in outcome 7, analysis 1]; GMR (Prior Alpha / Naïve Alpha) = 47.34 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 29: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; [p-value comment as in outcome 7, analysis 1]; GMR (Prior Alpha / Naïve Alpha) = 55.74 — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Number of Participants With Anti-CHIKV Total Antibody Titers of at Least 40,160 or 640
Description: Evaluation of Anti-CHIKV total antibody titer, as determined by immunoassay (ELISA), via proportion of participants with titers of at least 40, 160 or 640 on Days 1, 22, and 29.
Time Frame: Days 1, 22, and 29
Population: Immunogenicity evaluable population. 11 alphavirus naive participants were unable to attend their scheduled visit at Day 29.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Naive Alpha: All study participants received the same Investigational Product according to the same schedule. The alphavirus vaccine naïve participants served as controls.
Arm/Group | Experimental: Prior Alpha | Control: Naive Alpha
Number analyzed (Participants) | 30 | 30
Participants
  Day 1 Titers >=40 | 15 | 4
  Day 1 Titers >=160 | 4 | 1
  Day 1 Titers >=640 | 0 | 0
  Day 22 Titers >=40 | 30 | 30
  Day 22 Titers >=160 | 30 | 30
  Day 22 Titers >=640 | 30 | 26
  Day 29 Titers >=40: number analyzed (Participants) | 30 | 19
  Day 29 Titers >=40 | 30 | 19
  Day 29 Titers >=160: number analyzed (Participants) | 30 | 19
  Day 29 Titers >=160 | 30 | 19
  Day 29 Titers >=640: number analyzed (Participants) | 30 | 19
  Day 29 Titers >=640 | 30 | 17

9. Secondary Outcome: Percentage of Participants With 4-fold Rise in Anti-VEEV Neutralizing Antibody Response
Description: Evaluation of seroconversion rate of anti-VEEV neutralizing antibodies on Days 22 and 29 as determined by Plaque-Reduction Neutralization Test (PRNT80), where seroconversion is a 4-fold rise in titer over baseline.
Time Frame: Day 22 and 29
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Prior Alpha | Control: Naive Alpha
Number analyzed (Participants) | 30 | 30
percentage of participants
  Day 22 | 0 [0.0 to 11.4] | 0 [0.0 to 11.4]
  Day 29: number analyzed (Participants) | 30 | 19
  Day 29 | 0 [0.0 to 11.4] | 0 [0.0 to 16.8]
Statistical Analysis 1: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Test type: Superiority; p = 1.0000, Fisher Exact; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Test type: Superiority; p = 1.0000, Fisher Exact; [statistical method as in outcome 3, analysis 2]

10. Secondary Outcome: Percentage of Participants With Anti-VEEV PRNT Neutralizing Activity at or Above Selected Thresholds
Description: Evaluation of Anti-VEEV neutralizing antibody response, as determined by Plaque-Reduction Neutralization Test (PRNT80), via proportion of participants with titers of at least 40, 160 or 640 on Days 1, 22 and 29.
Time Frame: Day 1, 22, 29
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Prior Alpha | Control: Naive Alpha
Number analyzed (Participants) | 30 | 30
percentage of participants
  Day 1 (Titer >=40) | 90.0 [74.4 to 96.5] | 0 [0.0 to 11.4]
  Day 1 (Titer >=160) | 76.7 [59.1 to 88.2] | 0 [0.0 to 11.4]
  Day 1 (Titer >=640) | 53.3 [36.1 to 69.8] | 0.0 [0.0 to 11.4]
  Day 22 (Titer >=40) | 90.0 [74.4 to 96.5] | 0 [0.0 to 11.4]
  Day 22 (Titer >=160) | 80.0 [62.7 to 90.5] | 0 [0.0 to 11.4]
  Day 22 (Titer >=640) | 56.7 [39.2 to 72.6] | 0 [0.0 to 11.4]
  Day 29 (Titer >=40): number analyzed (Participants) | 30 | 19
  Day 29 (Titer >=40) | 90.0 [74.4 to 96.5] | 0 [0.0 to 16.8]
  Day 29 (Titer >=160): number analyzed (Participants) | 30 | 19
  Day 29 (Titer >=160) | 83.3 [66.4 to 92.7] | 0 [0.0 to 16.8]
  Day 29 (Titer >=640): number analyzed (Participants) | 30 | 19
  Day 29 (Titer >=640) | 60.0 [42.3 to 75.4] | 0 [0.0 to 16.8]
Statistical Analysis 1: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-VEEV PRNT neutralizing activity at or above selected thresholds by time point. Day 1: Subject with Titer >= 40; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-VEEV PRNT neutralizing activity at or above selected thresholds by time point. Day 1: Subject with Titer >= 160; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 3: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-VEEV PRNT neutralizing activity at or above selected thresholds by time point. Day 1: Subject with Titer >= 640; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 4: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-VEEV PRNT neutralizing activity at or above selected thresholds by time point. Day 22: Subject with Titer >= 40; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 5: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-VEEV PRNT neutralizing activity at or above selected thresholds by time point. Day 22: Subject with Titer >= 160; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 6: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-VEEV PRNT neutralizing activity at or above selected thresholds by time point. Day 22: Subject with Titer >=640; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 7: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-VEEV PRNT neutralizing activity at or above selected thresholds by time point. Day 29: Subject with Titer >= 40; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 8: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-VEEV PRNT neutralizing activity at or above selected thresholds by time point. Day 29: Subjects with Titer >= 160; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 9: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Null hypothesis for analysis of percentage of subjects with Anti-VEEV PRNT neutralizing activity at or above selected thresholds by time point. Day 29 : Subjects with Titer >=640; Test type: Superiority; p < 0.0001, Fisher Exact

11. Secondary Outcome: Geometric Mean Titer of Anti-VEEV Total Antibody Response
Description: Evaluation of Geometric Mean Titer of Anti-VEEV total antibody as determined by an immunoassay (ELISA) in prior alphavirus vaccine recipients versus alphavirus-naïve controls.
Time Frame: Day 1, 22, 29
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Experimental: Prior Alpha | Control: Naive Alpha
Number analyzed (Participants) | 30 | 30
titers
  Day 1 | 324.36 [195.37 to 538.52] | 14.03 [8.45 to 23.30]
  Day 22 | 2574.16 [1812.27 to 3656.35] | 14.92 [10.50 to 21.20]
  Day 29: number analyzed (Participants) | 30 | 19
  Day 29 | 2006.14 [1320.28 to 3048.31] | 16.94 [9.97 to 28.76]
Statistical Analysis 1: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 1: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 4]; GMR (Prior Alpha / Naïve Alpha) = 23.12, 95% CI 2-sided [11.54 to 46.35] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 22: Geometric mean ratio (prior alpha group over naïve alpha group) and 95% confidence interval; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 4]; GMR (Prior Alpha / Naïve Alpha) = 172.51, 95% CI 2-sided [106.60 to 279.19] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Day 29: Geometric mean ratio (prior alpha group over naive alpha group) and 95% confidence interval; Test type: Superiority; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 4]; GMR (Prior Alpha / Naïve Alpha) = 118.45, 95% CI 2-sided [61.76 to 227.16] — [estimate comment as in outcome 2, analysis 2]

12. Secondary Outcome: Percentage of Participants With 4-fold Rise in Total ELISA IgG Antibody Against VEEV
Description: Evaluation of seroconversion rate of Anti-VEEV total antibody, as determined by immunoassay (ELISA), on Days 22 and 29, where seroconversion is a 4-fold rise in titer over baseline.
Time Frame: Day 22, 29
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental: Prior Alpha | Control: Naive Alpha
Number analyzed (Participants) | 30 | 30
percentage of participants
  Day 22 | 86.7 [70.3 to 94.7] | 0 [0.0 to 11.4]
  Day 29: number analyzed (Participants) | 30 | 19
  Day 29 | 80.0 [62.7 to 90.5] | 0 [0.0 to 16.8]
Statistical Analysis 1: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Test type: Superiority; p < 0.0001, Fisher Exact; [statistical method as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Experimental: Prior Alpha vs Control: Naive Alpha; Test type: Superiority; p < 0.0001, Fisher Exact; Day 29 Note: A subject has a 4-fold rise at a visit if they achieve a titer at that visit that is at least 4-fold higher than their Day 1 titer

13. Secondary Outcome: Number of Participants With Anti-VEEV Total Antibody Titers of at Least 40,160 or 640
Description: Evaluation of Anti-VEEV total antibody titer, as determined by immunoassay (ELISA), via proportion of participants with titers of at least 40, 160, or 640 on Days 1, 22, and 29.
Time Frame: Days 1, 22, and 29
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Experimental : Prior Alpha: All study participants received the same Investigational Product according to the same schedule. Participants were prior recipients of experimental alphavirus vaccines.
Arm/Group | Experimental : Prior Alpha | Control: Naive Alpha
Number analyzed (Participants) | 30 | 30
Participants
  Day 1 Titers >=40 | 27 | 0
  Day 1 Titers >=160 | 23 | 0
  Day 1 Titers >=640 | 16 | 0
  Day 22 Titers >=40 | 27 | 0
  Day 22 Titers >=160 | 24 | 0
  Day 22 Titers >=640 | 17 | 0
  Day 29 Titers >=40: number analyzed (Participants) | 30 | 19
  Day 29 Titers >=40 | 27 | 0
  Day 29 Titers >=160: number analyzed (Participants) | 30 | 19
  Day 29 Titers >=160 | 25 | 0
  Day 29 Titers >=640: number analyzed (Participants) | 30 | 19
  Day 29 Titers >=640 | 18 | 0

ADVERSE EVENTS:
Time Frame: Local and systemic post-injection solicited events were collected through Day 8. Unsolicited adverse events were collected through Day 29. Serious adverse events and adverse events leading to withdrawal were collected through Day 183 end of study visit.
Arm/Group | Experimental : Prior Alpha | Control: Naive Alpha
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/30
Other Adverse Events (participants affected / at risk) | 17/30 | 17/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental : Prior Alpha (N=30) | Control: Naive Alpha (N=30)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental : Prior Alpha (N=30) | Control: Naive Alpha (N=30)
Injection site pain (General disorders) | 13 (13) | 9 (9)
Fatigue (General disorders) | 3 (3) | 3 (3)
Malaise (General disorders) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT03992872/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT03992872/SAP_003.pdf
  • Informed Consent Form (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT03992872/ICF_001.pdf